CLINICAL TRIAL: NCT04437901
Title: COVIDAR - International Registry on Arrhythmias in COVID-19
Brief Title: COVIDAR - Arrhythmias in COVID-19
Acronym: COVIDAR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Istituto Auxologico Italiano (Other); St George's University Hospitals NHS Foundation Trust (Other); University Hospital, Antwerp (Other); European Reference Network for Rare and Low Prevalence Complex Diseases of the Heart (ERN GUARDHEART) (Unknown); European Society of Cardiology (Network)
Responsible Party: Sponsor
Other Study IDs: HCB/2020/0333
Record Dates: First submitted 2020-05-28; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: COVID; Arrhythmia; Torsades de Pointe Caused by Drug; Qt Interval, Variation in; Atrioventricular Block; Atrial Fibrillation; Bradyarrhythmia; Ventricular Arrythmia
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrioventricular Block; Atrial Fibrillation; Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients: Patients admitted at one of the participating centres with highly suspected/confirmed infection with SARS-CoV-2.

SUMMARY:
BACKGROUND AND RATIONALE: There is very limited literature available on the arrhythmia occurrence in the context of an infection by the SARS-CoV2 virus. On the other hand, treatment strategies against the SARS-CoV2 virus may carry a risk of QTc prolongation and pro-arrhythmia/sudden death which may be amplified by concomitant use of other QTc-prolonging drugs and/or ion disbalances. COVIDAR is an international initiative to monitor the occurrence of arrhythmic events in the context of the SARS-CoV2 infection, to identify potential modifiable predisposing factors to reduce their incidence and to inform the best arrhythmia management options in this patient population.

MAIN OBJECTIVE: To describe the incidence and type of arrhythmic events in the context of the SARS-CoV2 infection.

STUDY DESIGN: patient registry (observational). Patients will not undergo any additional investigations. Only data that is generated during routine clinical care will be collected.

STUDY POPULATION: Patients admitted to the hospital highly suspected of or with confirmed COVID-19.

DETAILED DESCRIPTION:
The COVIDAR Registry is an international longitudinal multicentre observational study worldwide which aims to assess the incidence, type and risk factors of arrhythmias in the context of SARS-CoV2 infection, also providing relevant information on events/management and major cardiovascular outcomes. During the course of the registry patients will be followed up according to the usual practice of the centres. Drug prescriptions and indications to perform diagnostic/therapeutic procedures will be completely left to the treating physicians.

The registry population will consist of patients presenting with a suspicion of SARS-CoV2 infection, who are hospitalised in a medical or surgical department of the participating hospitals. Patients will officially be enrolled in the COVIDAR Registry if the COVID-19 disease has formally been noted or confirmed in the patient's medical record.

The registry will include all patients and collect data at the following timepoints:

* Admission: evaluation before SARS-CoV2 infection treatment initiation
* On-treatment: evaluation 24-28h after treatment initiation
* At any adverse event: evaluation if any adverse event occurs
* At discharge: evaluation of clinical status at the end of the admission period.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with highly suspected/confirmed infection with SARS-CoV-2.

Exclusion Criteria:

* Formal opposition by the patient to data collection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The registry population will consist of patients presenting with a suspicion of SARS-CoV2 infection, who are hospitalised in a medical or surgical department of the participating hospitals. Patients will officially be enrolled in the COVIDAR Registry if the COVID-19 disease has formally been noted or confirmed in the patient's medical record.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Arrhythmia | From date of admission until the date of first documented arrhythmic adverse event or date of death from any cause, whichever came first, assessed up to 12 months
  Any arrhythmic event occurring in COVID-19 patients during hospital admission:
  * Monomorphic ventricular tachycardia
  * Polymorphic ventricular tachycardia/Torsades de pointes (non-sustained)
  * Ventricular fibrillation
  * AV-block
  * Severe bradycardia, symptomatic and/or requiring treatment
  * New-onset atrial fibrillation
  * Other

SECONDARY OUTCOMES:
Electrocardiographic changes - Underlying rhythm | From date of admission until the date of first documented arrhythmic adverse event or date of death from any cause, whichever came first, assessed up to 12 months
  Categorical variable collecting the patient's underlying rhythm at baseline, on treatment and in case of arrhythmic adverse events): sinus rhythm, atrial fibrillation/flutter, other
Electrocardiographic changes - Atrioventricular conduction | From date of admission until the date of first documented arrhythmic adverse event or date of death from any cause, whichever came first, assessed up to 12 months
  Collected as a categorical (normal, 1st-, 2nd- or 3rd degree AV block) and a continuous (PR duration in ms) at baseline, on treatment and in case of arrhythmic adverse events)
Electrocardiographic changes - QRS duration | From date of admission until the date of first documented arrhythmic adverse event or date of death from any cause, whichever came first, assessed up to 12 months
  Collected as a continuous variable (ms) at baseline, on treatment and in case of arrhythmic adverse events)
Electrocardiographic changes - presence of Brugada QRS pattern | From date of admission until the date of first documented arrhythmic adverse event or date of death from any cause, whichever came first, assessed up to 12 months
  Collected as a categorical variable (not present, type 1 or type 2) at baseline, on treatment and in case of arrhythmic adverse events)
Electrocardiographic changes - QTc duration | From date of admission until the date of first documented arrhythmic adverse event or date of death from any cause, whichever came first, assessed up to 12 months
  Collected as a continuous variable (ms) at baseline, on treatment and in case of arrhythmic adverse events)
Laboratory abnormalities - electrolyte misbalance | From date of admission until the date of first documented arrhythmic adverse event or date of death from any cause, whichever came first, assessed up to 12 months
  Kalium, magnesium and calcium collected as continuous variables at baseline, on treatment and in case of arrhythmic adverse events). Will be reported as a categorical variable (presence/absence) of electrolyte misbalance
Laboratory abnormalities - cardiac biomarkers | From date of admission until the date of first documented arrhythmic adverse event or date of death from any cause, whichever came first, assessed up to 12 months
  Cardiac CK, troponin T and/or troponin I (where available) collected as a continuous variable at baseline, on treatment and in case of arrhythmic adverse events)
Laboratory abnormalities - renal function | From date of admission until the date of first documented arrhythmic adverse event or date of death from any cause, whichever came first, assessed up to 12 months
  Creatinine clearance at baseline, on treatment and in case of arrhythmic adverse events)
Laboratory abnormalities - liver function | From date of admission until the date of first documented arrhythmic adverse event or date of death from any cause, whichever came first, assessed up to 12 months
  Liver enzymes collected at at baseline, on treatment and in case of arrhythmic adverse events)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Arbelo, MD, PhD, MSc, Study Chair — Hospital Clinic of Barcelona; Arthur A Wilde, MD, PhD, Study Director — Amsterdam UMC; Lia Crotti, MD, PhD, Study Director — Istituto Auxologico Italiano, IRCCS; Elijah Behr, MD, PhD, Study Director — St George's University Hospitals NHS Foundation Trust; Hein Heidbuchel, MD, PhD, Study Director — University Hospital, Antwerp
Locations (5):
- Antwerp University Hospital, Antwerp, Belgium
- Istituto Auxologico Italiano, IRCCS, Milan, Italy
- Amsterdam UMC, Amsterdam, AZ, Netherlands
- Hospital Clinic of Barcelona, Barcelona, Spain
- St. Georges University Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided